CLINICAL TRIAL: NCT05723133
Title: A Randomized Controlled Trial Comparing Manual Versus Powered Toothbrushes With Visual Feedback
Brief Title: Visual Feedback on Brushing Technique and Habits on Patient Oral Hygiene
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BC-11037
Record Dates: First submitted 2023-01-30; First posted 2023-02-10 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Toothbrushing; Oral Hygiene; Dental Plaque
Keywords: Dental plaque; Toothbrush; Oscillating-rotating; Manual; Electric; Dental Plaque Index; Electrical Equipment and Supplies
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial with 3 treatment arms (control group: manual toothbrush; test group 1: electric toothbrush without digital visual feedback; test group 2: electric toothbrush with visual feedback). Every patient received the same initial treatment and oral hygiene instructions. Sealed envelops will determine in which group the patient will participate.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The patient and treating dentist cannot be masked. The investigators and outcome assessors are masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active Comparator: Control group: Manual Toothbrush (Active Comparator): Patients will receive oral hygiene instructions and a new manual toothbrush
  Interventions: Behavioral: Oral hygiene instructions
- Test group: Electric Toothbrush without visual feedback (Experimental): Patients will receive the same oral hygiene instructions and an electric toothbrush without daily personal feedback using the brushing application.
  Interventions: Device: Electric toothbrush; Behavioral: Oral hygiene instructions
- Test group: Electric Toothbrush with visual feedback (Experimental): Patients will receive the same oral hygiene instructions and an electric toothbrush with daily personal feedback using the brushing app (Oral-B app).
  Interventions: Device: Electric toothbrush; Behavioral: Oral hygiene instructions

INTERVENTIONS:
Device: Electric toothbrush — Patients will receive oral hygiene instructions and an electric toothbrush with or without daily personal feedback using the brushing app (Oral-B app).
  Arms: Test group: Electric Toothbrush with visual feedback; Test group: Electric Toothbrush without visual feedback
Behavioral: Oral hygiene instructions — The same oral hygiene instructions are given to all patients. It is important for the patient to scrupulously follow these oral hygiene instructions at home and carry them out daily.

SUMMARY:
The goal of this clinical trial is to learn about the influence of providing visual feedback on brushing technique and habits on oral health of patients undergoing periodontal treatment.

The main question[s] it aims to answer are:

* Is patients' oral health improved by providing visual feedback on their brushing technique using the smartphone brushing app?
* Is there behavioural change of patients based on this daily visual feedback? Participants will receive oral hygiene instructions after initial periodontal treatment and will be randomized in group 1, 2 or 3. Participants will be asked to

  * fulfill a brushing diary with the time of brushing every day.
  * come back for a check-up appointment every 3 weeks during the study to evaluate oral hygiene.

Researchers will compare manual toothbrush, electric toothbrush without daily personal feedback and electric toothbrush with daily personal feedback to see if visual feedback provide improved oral health

DETAILED DESCRIPTION:
Periodontitis is gum disease with jawbone deterioration. Diagnosis is based on clinical examination: plaque score, pocket measurement (measuring the pockets or gum pockets around the teeth with a probe), gingival bleeding index (= bleeding after probing) and radiographic examination. Smoking, genetic factors, and systemic diseases such as diabetes, for example, are known risk factors for this condition. Treatment consists of a deep cleaning, where the tooth roots are freed of plaque and tartar under local anaesthesia, complemented by the necessary oral hygiene instructions. It is important that patients follow these oral hygiene instructions carefully at home and perform them daily, as the aim is to achieve optimal oral hygiene. Good oral hygiene is fundamental in the treatment of periodontitis (Arweiler et al, 2018).

Despite many patients undergoing the proposed professional treatment (deep cleaning), they are often insufficiently able to remove the dental plaque present on a daily basis. To optimise brushing efficiency, both behavioural change and improved brushing technique should be obtained at the patient level.

The primary aim of this randomised clinical trial is to improve patients' oral health by providing visual feedback on their brushing technique using the smartphone brushing app. The secondary aim of the study is to investigate possible behavioural changes of patients based on this daily visual feedback.

Patients requiring periodontal treatment will be recruited at the Department of Periodontology & Oral Implantology at Ghent University Hospital. Patients will be assigned to three groups by randomisation. In group 1, patients will receive oral hygiene instructions and a new manual toothbrush. In group 2, patients receive the same oral hygiene instructions and a basic electric toothbrush without daily personal feedback using the brushing application. In group 3, patients receive the same oral hygiene instructions and an electric toothbrush with daily personal feedback using the brushing app (Oral-B app). No raw study data will be transferred to Oral B. The only data that will be available to Oral-B is the data that will be included in the publication of this study (A1 article). The use of the app does not require registration of personal data. Brushing time, tooth surface cleaning and brushing pressure will be recorded. Patients will only complete the brushing time in the brushing diary.

Oral hygiene will be evaluated at the start and every 3 weeks during the study through a check-up appointment. Only the first (after 3 weeks) and the last check-up appointment (after 12 weeks) are standard protocol, the remaining appointments (after 6 and 9 weeks) are study-specific. Oral hygiene will be assessed by: plaque score, gingival bleeding index, brushing frequency and brushing duration. The full study will take 12 weeks. Pocket depth will be measured according to usual protocols, namely at intake and at the last check-up (after 12 weeks). The patient's brushing technique and frequency will be recorded through a brushing diary completed by the patient. Where necessary, oral hygiene can be adjusted during each sitting. The check-up after 3 weeks and 12 weeks with measurement of plaque scores, gingival bleeding index and pocket depth are part of the standard protocol for treating periodontitis and are therefore not study-specific. Monitoring after 6 and 9 weeks are study-specific. The primary goal will be evaluated by comparing plaque scores and gingival bleeding index at intake with those at the final check. The secondary goal will be evaluated by brushing frequency and brushing duration throughout the study course. All data collected will be pseudonymised.

Overview:

* Consultation 1 - at start:

  o Standard treatment: Evaluation of oral hygiene Determination of clinical score: plaque score, gingival bleeding index Determination of pocket depth

  o Study-specific treatment (duration: 10 minutes): Clinical photographs
* Consultation 2 - after 3 weeks:

  o Standard treatment: Evaluation of oral hygiene and brushing frequency. Determination of clinical score: plaque score, gingival bleeding index

  o Study-specific treatment (duration: 10 minutes): Clinical photographs
* Consultation 3 - after 6 weeks:

  o Study-specific treatment (duration: 30 minutes ): Evaluation of oral hygiene + clinical photographs Determination of clinical score: plaque score, gingival bleeding index
* Consultation 4 - after 9 weeks:

  o Study-specific treatment (duration: 30 minutes ): Evaluation of oral hygiene + clinical photographs Determination of clinical score: plaque score, gingival bleeding index
* Consultation 5 - after 12 weeks:

  o Standard treatment: Evaluation of oral hygiene and brushing frequency. Determination of clinical score: plaque score, gingival bleeding index Determination of pocket depth

  o Study-specific treatment (duration: 10 minutes): Clinical photographs
* Completion of the brushing diary by the patient:

  * Brushing time, cleaning of tooth surfaces, brushing pressure, brushing technique, frequency and motivation
  * 2x a day, 2 min per brushing

ELIGIBILITY:
Inclusion Criteria:

* Patients in need of periodontal treatment
* Willing to keep a brushing diary
* Possess a smartphone so that they are able to install and handle the application on their phone

Exclusion Criteria:

* Smoking
* Systemic disease
* Pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-02-24 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Oral hygiene with or without visual feedback | 12 weeks
  Comparing the plaque scores at intake with those at final check-up
Oral hygiene with or without visual feedback | 12 weeks
  Comparing the gingival bleeding index at intake with those at final check-up

SECONDARY OUTCOMES:
Behavioural changes | 12 weeks
  Brushing frequency will be evaluated using the brushing diary (minutes)
Behavioural changes | 12 weeks
  Brushing durations will be evaluated using the brushing diary (number of times)

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Christiaens, Prof. Dr., Principal Investigator — University Ghent
Locations (4):
- Belgium (4):
  - BV Paro Glibert, Geraardsbergen, Oost-Vlaanderen
  - Ghent University, Ghent, Oost-Vlaanderen
  - Praktijk voor Parodontologie, Sint-Niklaas, Oost-Vlaanderen
  - Centrum voor Parodontologie en Orale Implantologie, Zottegem, Oost-Vlaanderen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Adam R, Ram Goyal C, Qaqish J, Grender J. Evaluation of an oscillating-rotating toothbrush with micro-vibrations versus a sonic toothbrush for the reduction of plaque and gingivitis: results from a randomized controlled trial. Int Dent J. 2020 Apr;70 Suppl 1(Suppl 1):S16-S21. doi: 10.1111/idj.12569. PMID 32243576
- [Result] Nathoo S, Mankodi S, Mateo LR, Chaknis P, Panagakos F. A clinical study comparing the supragingival plaque and gingivitis efficacy of a specially engineered sonic powered toothbrush with unique sensing and control technologies to a commercially available manual flat-trim toothbrush. J Clin Dent. 2012;23 Spec No A:A11-6. PMID 23448083
- [Result] Grender J, Ram Goyal C, Qaqish J, Adam R. An 8-week randomized controlled trial comparing the effect of a novel oscillating-rotating toothbrush versus a manual toothbrush on plaque and gingivitis. Int Dent J. 2020 Apr;70 Suppl 1(Suppl 1):S7-S15. doi: 10.1111/idj.12571. PMID 32243573